CLINICAL TRIAL: NCT03448926
Title: A Prospective Registry Study to Evaluate the Effect of the DCISionRT Test on Treatment Decisions in Patients with DCIS Following Breast Conserving Therapy
Brief Title: The PREDICT Registry:
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: PreludeDx (Industry)
Responsible Party: Sponsor
Other Study IDs: Ext00000206
Record Dates: First submitted 2018-02-16; First posted 2018-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: DCIS
Keywords: DCIS; molecular testing; risk of recurrence; treatment decision; decision impact; predictive
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — primary tumor blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- DCIS: Patients must have histologically confirmed ductal carcinoma in situ (DCIS) in a single breast without evidence of invasive cancer (presence of lobular carcinoma in situ (LCIS) or other benign breast disease in addition to DCIS is acceptable)
  Interventions: Other: Treatment Recommendation Surveys; Device: 7-gene biosignature

INTERVENTIONS:
Other: Treatment Recommendation Surveys — Treatment Recommendation Surveys are completed by the treating physicians before and after receiving results from the DCISionRT test, which is prognostic for risk of recurrence over 10 years and predictive for benefit from radiation therapy.
Device: 7-gene biosignature — Ordering the 7-gene biosignature assay (DCISionRT) as a part of routine care for DCIS is a prerequisite (inclusion criterion) for the study. The study is not designed to determine the efficacy of the assay, rather it is designed to meausre the impact of the assay results on treatment decisions for patients with DCIS.

SUMMARY:
This is a prospective, non-interventional (observational) cohort study conducted within the medical network of the participating investigators and institutions. Patients meeting the eligibility criteria (see below) will be eligible for participation and the investigators will obtain written informed consent. A central Institutional Review Board (IRB), WCG IRB, will approve the protocol and each participating institution.

DETAILED DESCRIPTION:
After a diagnosis of DCIS, the most representative tissue block (or 10 sections mounted on charged slides cut at 3-4 microns) will be sent to PreludeDx for DCISionRT. The most representative specimen should be selected from tissue collected via direct tumor biopsy (either core needle or excisional biopsy) as part of routine patient care. Patients must be enrolled in the study and the enrollment and pre-testing data forms must be completed and submitted before the DCISionRT results are reported. Then, after review of the DCISionRT results, the investigators complete and submit the post-testing data form. The patient may then be followed for up to 10 years (or until death) with completion of 5- and 10-year follow-up forms.

All study data will be stored in an encrypted, HIPAA-compliant database maintained by the coordinating center. Each consented patient will be assigned a unique Study ID number. Study personnel at each institution will maintain an electronic key to link the Study IDs of its own patients to the patients' local medical record number. All personal health information (PHI) will remain at the local institution and only de-identified data will be uploaded to the national registry. No genetic test results that may be used to identify the patient will be included in the database.

This study is designed to assess the magnitude of and conditions impacting physician treatment recommendations based on the DCISionRT test results, assessing patient preference, and within various clinicopathologic subgroups. This will also be the largest prospective determination of IBR outcomes with DCISionRT test result correlates to date.

Part I of the PREDICT Registry recently completed enrollment of 2,500 subjects for whom DCISionRT results had been reported using the original test protocol that classified patients into two risk groups, Low Risk and Elevated Risk.64

Part II of the PREDICT Registry will enroll up to an additional 3,000 subjects from 15 to 30 sites within the United States with each site enrolling between 100 and 300 patients. DCISionRT results will be reported using the updated test protocol that classifies patients into three risk groups, Low Risk, Elevated Risk and Residual Risk. Part II study procedures will be conducted exactly the same as Part I, except that further patient demographics and treatment preference, treatment recommendation details, and patient upstaging will be collected. Additional questions will be asked to determine how physicians use the Residual Risk group classification to make treatment decisions. De-identified imaging data may also be collected, and de-identified patient tissue samples may be collected after 1 year.

ELIGIBILITY:
Inclusion criteria

1. Patient must have histologically confirmed ductal carcinoma in situ (DCIS) in a single breast (presence of lobular carcinoma in situ (LCIS) or other benign breast disease in addition to DCIS is acceptable).
2. Patient must have the DCISionRT test ordered during routine patient care.
3. Patient must be eligible for or have recently completed breast conserving surgery.
4. Patient must be eligible to receive radiation and/or systemic treatment.
5. Patient must be 30 to 85 years old.
6. Patient must have tumor size of less than 6 cm.
7. Patient must have been diagnosed with DCIS within 120 days of consent.

Exclusion criteria

1. Patient tissue is insufficient to generate DCISionRT test results or required DCISionRT inputs (age, tumor size, margin status, palpability) are missing.
2. Patient has evidence of invasive breast cancer, including microinvasion, lymph node involvement, or Paget's disease of the nipple or suspicious mammogram findings in the lymph nodes or contralateral breast.
3. Patient has been surgically treated with an ipsilateral mastectomy for primary DCIS.
4. Patient has had any prior ipsilateral or contralateral breast DCIS or invasive breast cancer.
5. Patient has a prior history of in-field radiation in the ipsilateral breast.
6. Patient has had prior systemic endocrine or chemotherapy prior to testing.
7. Patient is pregnant.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the clinical practices of the participating investigators and institutions. Patients who have been recently diagnosed with DCIS and are being evaluated for the need for further therapy will be screened for eligibility per the following eligibility criteria. Female patients 30 to 85 years with histologically confirmed ductal carcinoma in situ (DCIS) in a single breast of size less than 6 cm without evidence of invasive or microinvasive cancer and clinically eligible to receive breast-conserving surgery with or without radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Percent of Cases with Changes in Treatment Recommendation | From enrollment to the beginning of treatment.
  The percent of cases in which treatment recommendations are changed after the test DCISionRT test results become available. The study will collect details on physician treatment recommendations and patient preference before and after the availability of the molecular test (DCISionRT) results. The data elements include type of surgery (lumpectomy, therapeutic mastectomy, contralateral prophylactic mastectomy), type of radiation therapy (none, IORT, APBI/PBI, whole breast RT, boost) and endocrine therapy.

SECONDARY OUTCOMES:
Function of Tumor Factors | 5 years
  Percent of patients for which the recommended treatments change after DCISionRT results are known as a function of tumor factors (tumor size, grade, architecture, necrosis, palpability, surgical margins, hormone receptor status).
Function of Tumor and Demographic Factors | From enrollment to the beginning of treatment.
  Percent of patients for which the recommended treatments change after DCISionRT results are known as a function of tumor factors (tumor size, nuclear grade, architecture, necrosis, palpability, surgical margins, hormone receptor status).
  Percent of patients for which the recommended treatments change after DCISionRT results are known as a function of demographic factors (age; ethnicity; family history, education, marital status, geographic region).

OTHER OUTCOMES:
Distribution of DCISionRT scores across the cohort | From enrollment to the beginning of treatment.
  Each patient will receive the following results from the DCISionRT test: Decision Score (DS, 0.8-10.0), Residual Risk subtype (DS 9.2).
Function of Geographic Region | From enrollment to the beginning of treatment.
  Percent of patients for which the recommended treatments change after DCISionRT results are known as a function of the geographic region of the investigator, type of institution, or type of treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Bremer, PhD, Principal Investigator — PreludeDx; Pat W Whitworth, MD, Study Chair — PreludeDx; Rachel Rabinovitch, MD, Study Chair — University of Colorado, Denver; Pat Borgen, MD, Study Chair — Maimonides Medical Center
Locations (15):
- United States (15):
  - Arizona Center for Cancer Care, Phoenix, Arizona
  - Sutter Institute for Medical Research, Sacramento, California
  - Mills-Peninsula Medical Center, San Mateo, California
  - University of Colorado Denver, Aurora, Colorado
  - UC Health - Memorial Hospital, Colorado Springs, Colorado Springs, Colorado
  - St. Joseph's Hospital Tampa, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Comprehensive Breast Care, Troy, Michigan
  - Maimonides Cancer Center, Brooklyn, New York
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Nashville Breast Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah C, Whitworth P, Vicini FA, Narod S, Gerber N, Jhawar SR, King TA, Mittendorf EA, Willey SC, Rabinovich R, Gold L, Brown E, Patel A, Vargo J, Barry PN, Rock D, Friedman N, Bedi G, Templeton S, Brown S, Gabordi R, Riley L, Lee L, Baron P, Majithia L, Mirabeau-Beale KL, Reid VJ, Hirsch A, Hwang C, Pellicane J, Maganini R, Khan S, MacDermed DM, Small W, Mittal K, Borgen P, Cox C, Shivers SC, Bremer T. The Clinical Utility of a 7-Gene Biosignature on Radiation Therapy Decision Making in Patients with Ductal Carcinoma In Situ Following Breast-Conserving Surgery: An Updated Analysis of the DCISionRT(R) PREDICT Study. Ann Surg Oncol. 2024 Sep;31(9):5919-5928. doi: 10.1245/s10434-024-15566-5. Epub 2024 Jun 25. PMID 38916700
- [Background] Dabbs D, Mittal K, Heineman S, Whitworth P, Shah C, Savala J, Shivers SC, Bremer T. Analytical validation of the 7-gene biosignature for prediction of recurrence risk and radiation therapy benefit for breast ductal carcinoma in situ. Front Oncol. 2023 May 19;13:1069059. doi: 10.3389/fonc.2023.1069059. eCollection 2023. PMID 37274253
- [Background] Vicini FA, Mann GB, Shah C, Weinmann S, Leo MC, Whitworth P, Rabinovitch R, Torres MA, Margenthaler JA, Dabbs D, Savala J, Shivers SC, Mittal K, Warnberg F, Bremer T. A Novel Biosignature Identifies Patients With DCIS With High Risk of Local Recurrence After Breast Conserving Surgery and Radiation Therapy. Int J Radiat Oncol Biol Phys. 2023 Jan 1;115(1):93-102. doi: 10.1016/j.ijrobp.2022.06.072. Epub 2022 Sep 15. PMID 36115740
- [Background] Warnberg F, Karlsson P, Holmberg E, Sandelin K, Whitworth PW, Savala J, Barry T, Leesman G, Linke SP, Shivers SC, Vicini F, Shah C, Weinmann S, Mann GB, Bremer T. Prognostic Risk Assessment and Prediction of Radiotherapy Benefit for Women with Ductal Carcinoma In Situ (DCIS) of the Breast, in a Randomized Clinical Trial (SweDCIS). Cancers (Basel). 2021 Dec 3;13(23):6103. doi: 10.3390/cancers13236103. PMID 34885211
- [Background] Shah C, Bremer T, Cox C, Whitworth P, Patel R, Patel A, Brown E, Gold L, Rock D, Riley L, Kesslering C, Brown S, Gabordi R, Pellicane J, Rabinovich R, Khan S, Templeton S, Majithia L, Willey SC, Warnberg F, Gerber NK, Shivers S, Vicini FA. Correction to: The Clinical Utility of DCISionRT(R) on Radiation Therapy Decision Making in Patients with Ductal Carcinoma In Situ Following Breast-Conserving Surgery. Ann Surg Oncol. 2021 Dec;28(Suppl 3):878. doi: 10.1245/s10434-021-10138-3. No abstract available. PMID 33997922